CLINICAL TRIAL: NCT03058549
Title: Family Expectations: Impact Evaluation of Program for Expectant Couples
Brief Title: Impact Evaluation of Family Expectations: A Program to Strengthen the Relationships of Disadvantaged Expectant Couples
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Strategies (Other)
Collaborators: Children's Bureau - Administration for Children and Families (Other); University of Denver (Other)
Responsible Party: Principal Investigator, Galena Rhoades, Prinicipal Investigator, University of Denver
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 860135
Record Dates: First submitted 2017-02-10; First posted 2017-02-23 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Committed Couple Expecting a Child; Parenting; Family Relations
Keywords: Expectant parents; Relationship education

STUDY DESIGN:
Masking Description: Open Label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Family Expectations (Experimental): Family Expectations includes 36 hours of relationship education and parenting content, coaching sessions for couples, and group case management/referral information about local resources. Each couple will also complete an initial case management assessment, followed by referrals to any needed services, such as employment, substance abuse, mental health, housing, etc. Based on need, couples will have the option of additional case management/coaching services during their involvement in Family Expectations.
  Interventions: Behavioral: Family Expectations
- Control Group (No Intervention): The control group will not receive the intervention though they are able to seek and obtain any services they wish in the community (Treatment as Usual).

INTERVENTIONS:
Behavioral: Family Expectations — Relationship education and referral services for expectant couples.
  Arms: Intervention: Family Expectations

SUMMARY:
This study investigates the effectiveness of a program to strengthen the relationships of disadvantaged expectant couples, and to increase co-parenting, father involvement, and economic stability. Couples are randomly assigned to Family Expectations or a control group, and assessed at baseline and one year.

DETAILED DESCRIPTION:
The birth of a child can trigger relationship distress and dissolution. Family Expectations (FE) targets the transition to parenthood as a critical time to help couples focus on family success. Regardless of whether couples are married or unmarried, the goal of FE is to strengthen relationships and advance the well-being of economically disadvantaged couples who are expecting a baby or who are new parents, and to improve the lives of their children. The FE program, including the Becoming Parents (BP) curriculum and supplemental services, is designed to address specific risk factors that affect individual family members and the relationships among them, and to build protective factors that help families avoid, minimize, or manage risks (e.g., individual maladaptation [mother, father, child], couple relationship difficulties, parenting difficulties, and economic insufficiency).

A total of 1,355 couples will be randomly assigned to either Family Expectations (n = 813; 60%) or an untreated control group (n = 542; 40%). Once assigned, participants in the study will complete baseline questions by survey. Those assigned to the FE track will be scheduled for services with the FE intervention team and the control group will not receive the FE intervention. Members of the intervention and control groups will be surveyed both before they are randomly assigned and 12 months later. The study will examine if the Family Expectations program is associated with improved outcomes on relationship quality, stability, parenting quality, father involvement, child wellbeing, and hopefulness about employment.

ELIGIBILITY:
Inclusion Criteria:

1. Both partners are willing to participate
2. Partners have a commitment to be together as a couple
3. Both partners are the biological parents of a child in a current pregnancy or of a child born within the past 3 months
4. Fluent in English (study and intervention materials are in English)

Exclusion Criteria:

1. Either or both partners have taken part in Family Expectations services before

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2640 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Relationship adjustment | Baseline and 1 year post baseline (to assess change over time). Change (or maintenance) relative to control group will be assessed across the two time points.
  This outcome will be measured by a composite of measures to relationship quality (support and affection, global relationship satisfaction, and confidence in the future of the relationship). Respondents will self-report using survey methods.
Relationship stability | 1 year post baseline
  Couple remains romantically involved. Self-reported by survey methods.
Individual wellbeing | Baseline and 1 year post baseline. Change (or maintenance) relative to control group will be assessed across the two time points.
  Symptoms of depression and anxiety. Respondents will self-report using survey methods.
Co-parenting quality | 1 year post baseline.
  The quality of the co-parenting relationship between the expectant partners will be self-reported using survey methods.
Child outcomes | 1 year post baseline.
  Infant temperament and wellbeing will be assessed by parent self-report using survey methods.
Interaction quality | Baseline and 1 year post baseline. Change (or maintenance) relative to control group will be assessed across the two time points.
  This outcome will be measured by a composite of measures that assess communication and conflict management abilities (communication skills, constructive conflict management, destructive conflict management). Respondents will self-report using survey methods.

SECONDARY OUTCOMES:
Changes in Income | Baseline and 1 year post baseline. Change relative to control group will be assessed across the two time points.
  Income will be measured by self-report using survey methods.

CONTACTS AND LOCATIONS:
Overall Officials: Galena K Rhoades, Ph.D., Principal Investigator — University of Denver
Locations (1):
- Public Strategies, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided